CLINICAL TRIAL: NCT04690205
Title: Hospital-at-Home Care Model to Optimize End-of-Life (EOL) Care for Patients With Hematologic Malignancies: A Pilot Feasibility Study
Brief Title: Hospital at Home at EOL in Heme Malignancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Medically Home (Unknown)
Responsible Party: Principal Investigator, El-Jawahri, Areej,M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-468
Record Dates: First submitted 2020-12-26; First posted 2020-12-30 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Hematologic Malignancy
Keywords: Hematologic Malignancy; Home Care Services
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Death Domain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- End of Life (EOL) Care at at Home (Experimental): End of Life (EOL) Care at at Home intervention entails the following: patient-reported symptoms and home monitored vital signs and body weight with appropriate triggers for phone calls and home visits, and regular communication with oncology clinicians regarding care delivered at home to ensure continuity of care.
  Interventions: Other: End of Life (EOL) Care at at Home

INTERVENTIONS:
Other: End of Life (EOL) Care at at Home — Remote monitoring and home-based care designed for patients with advanced hematologic malignancies

SUMMARY:
This study is evaluating an intervention, which the investigators call "Optimize End of Life (EOL) Care at Home," that entails remote patient monitoring and home-based supportive care for patients with advanced hematologic malignancies.

DETAILED DESCRIPTION:
This research study is a single arm pilot feasibility study, which is the first-time investigators are examining this care at home intervention in patients with advanced hematologic malignancies.

The research study procedures include screening for eligibility, questionnaires, remote patient monitoring (e.g. patient-reported symptoms, home monitored vital signs) and hospital care at home (e.g. providing maximal supportive care to to address and manage patients' symptoms) and structured communications oncology clinicians to optimize end of life care for patients with advanced hematologic malignancies.

Participants will include 3 groups:

1) Enrolled patients with advanced hematologic malignancies receiving the end of life (EOL) care at home intervention; 2) caregivers of these patients; and 3) oncology clinicians caring for these patients.

Participants will be in this research study for approximately six months after consent. It is expected that about 30 patients, 30 caregivers, and 15 oncology clinicians will take part in this research study.

Medically Home company is supporting this research study by providing funding.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* diagnosed with relapsed or refractory hematologic malignancy
* must be receiving treatment with non-curative intent or supportive care alone based on the intent of chemotherapy as reported in order entry or Electronic Health Record
* deemed eligible to receive EOL care at home based on the primary oncologist's assessment
* Able to communicate and respond to questionnaires in English or with the assistance of an interpreter.
* residing within 50 miles of MGH. Of note, patients requiring supportive transfusions in the oncology clinic will still be eligible to participate.

Exclusion Criteria:

* Those with uncontrolled psychiatric illness or impaired cognition interfering with their ability to understand study procedures and provide written informed consent as determined by the primary oncologist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Enrollment Rate | 6 months
  The primary endpoint is feasibility. The proposed intervention will be deemed feasible if at least 60% (95% confidence interval +/- 18%) of eligible patients are enrolled in the study.
Retention Rate | 6 months
  The primary endpoint is feasibility. The proposed intervention will be deemed feasible if at least 80% of enrolled participants will complete a minimum of 60% of their daily assessments (i.e. patient-reported symptoms)

SECONDARY OUTCOMES:
Acceptability of the intervention | 6 months
  Qualitative acceptability ratings from patients, caregivers, and oncology clinicians defined by perceptions of usefulness, effectiveness, and relevance of the intervention obtained via interviews regarding acceptability from patients, family caregivers, and oncology clinicians.
Patient Quality of Life (Functional Assessment of Cancer Therapy-General - Fact-G) | up to 6 months
  Change in quality of life as measured by the FACT-G throughout the study. FACT-G score ranges from 0 to 108 points with higher score indicating better quality of life
Caregiver Quality of Life (CareGiver Oncology QOL) | 6 months
  Change in caregiver quality of life as measured by the CarGOQOL throughout the study. Caregiver Oncology QOL questionnaire ranges from 0 to 100 points with higher scores indicating better caregiver quality of life
Patient Symptom Burden (using the Edmonton Symptom Assessment Scale-revise) | up to 6 months
  Change in patient symptom burden measured with Edmonton Symptom Assessment System-revised (ESAS-r). Scores range from 0-100 with higher scores indicate worse symptom burden.
Caregiver Burden | up to 6 months
  Caregiving burden will be assessed using the Caregiver Reaction Assessment (CRA) caregiving burden. The CRA score ranges from 24-120, with higher score indicating higher caregiving burden
Health Care Utilization | 6 months
  Electronic Health Records (EHR) will be used to assess patient health care utilization including hospitalizations, chemotherapy use, and emergency department visits at the end of life.
Patient psychological distress (using the Hospital Anxiety and Depression Scale (HADS)) | Up to 6 months
  The Hospital Anxiety and Depression Scale (HADS) will be used to assess patient psychological distress. The HADS score ranges from 0-21 with higher score indicating more psychological distress.
Caregiver psychological distress (using the Hospital Anxiety and Depression Scale (HADS)) | Up to 6 months
  The Hospital Anxiety and Depression Scale (HADS) will be used to caregiver psychological distress. The HADS score range from 0-21 with higher scores indicating worse psychological distress
Caregiver Satisfaction with patient's end of life (EOL) care using the FAMCARE | Up to 6 months
  Nine items from the FAMCARE will be used to assess caregivers' satisfaction with the quality of medical services provided to them and the patient at the end of life. FAMCARE provides rating of quality of death on a scale of 0-10, with higher scores indicating best possible death. FAMCARE also provides a total score ranges 0-24, with higher score indicating better satisfaction with EOL care

CONTACTS AND LOCATIONS:
Overall Officials: Areej El-Jawahri, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] Nipp RD, Shulman E, Smith M, Brown PMC, Johnson PC, Gaufberg E, Vyas C, Qian CL, Neckermann I, Hornstein SB, Reynolds MJ, Greer J, Temel JS, El-Jawahri A. Supportive oncology care at home interventions: protocols for clinical trials to shift the paradigm of care for patients with cancer. BMC Cancer. 2022 Apr 9;22(1):383. doi: 10.1186/s12885-022-09461-z. PMID 35397575